CLINICAL TRIAL: NCT04617509
Title: An Open, One-sequence, Three-period Study in Healthy Subjects to Evaluate Pharmacokinetics and Food Effect After Oral Single Dosing of Two Different Solid Formulations of GS-248
Brief Title: A Study in Healthy Subjects to Evaluate Pharmacokinetics and Food Effect After Dosing of GS-248
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gesynta Pharma AB (Industry)
Collaborators: CTC Clinical Trial Consultants AB (Industry); Research Institutes of Sweden (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GS-1002
Record Dates: First submitted 2020-05-27; First posted 2020-11-05 (Actual); Results first posted 2021-08-31 (Actual); Last update posted 2021-08-31 (Actual); Status verified 2021-08

CONDITIONS: Pharmacokinetic
Keywords: Pharmacokinetic

STUDY DESIGN:
Intervention Model Description: The study is divided in two parts. Part I will evaluate PK, safety and tolerability of a single oral dose of two different formulations of GS-248 in fasting conditions. Part II will evaluate PK, safety and tolerability of one of the two different formulations of GS-248 in fed conditions. Subjects are expected to participate in both Part I and Part II.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Part I GS-248 Formulation A (Experimental): Formulation A given in fasting state.
  Interventions: Drug: Formulation A GS-248
- Part I GS-248 Formulation B (Active Comparator): Formulation B given in fasting state.
  Interventions: Drug: Formulation B GS-248
- Part II GS-248 Formulation A or B (Other): Formulation A or B given in fed condition
  Interventions: Drug: Formulation A GS-248; Drug: Formulation B GS-248

INTERVENTIONS:
Drug: Formulation A GS-248 — Formulation A of GS-248 in a capsule, dose 120 mg given as a single-dose of 3 capsules a´40 mg.
  Arms: Part I GS-248 Formulation A; Part II GS-248 Formulation A or B
Drug: Formulation B GS-248 — Formulation B of GS-248 in a capsule, dose 120 mg given as a single-dose of 3 capsules a´40 mg.
  Arms: Part I GS-248 Formulation B; Part II GS-248 Formulation A or B

SUMMARY:
The study will collect information about pharmacokinetics (PK), safety and tolerability following a single dose of GS-248 in two different oral solid formulations in capsules to healthy subjects. It will also collect information about pharmacokinetics (PK), safety and tolerability following a single dose of one of the two formulations of GS-248 in fed condition.

DETAILED DESCRIPTION:
The study is divided in two parts. Part I will evaluate PK, safety and tolerability of a single oral dose of two different formulations of GS-248 in fasting conditions. Part II will evaluate PK, safety and tolerability of one of the two different formulations of GS-248 in fed conditions.

In Part I, a single oral dose of GS-248 in two different solid formulations will be administered to 14 healthy subjects. All subjects will first receive Formulation A and then Formulation B. A wash-out period of at least 4 days will be applied between the IMP administrations. Both doses contain 120 mg GS 248. For Part I, subjects will come to the clinic for single dose administration of Formulation A or Formulation B, respectively, and PK and safety assessments. Safety assessments include AE reporting, physical examination, ECG, vital signs, body temperature, and blood sampling for analysis of safety laboratory parameters.

After evaluation of the PK profiles of Formulation A and B in Part I of the study, one formulation will be selected to be given following intake of a standardised breakfast in Part II of the study. Subjects will return to the clinic for a second dose of the selected formulation, yet now in fed conditions. The assessments during fed conditions will be the same as during fasting conditions except that the subjects will consume a high-fat high-calorie breakfast 30 minutes prior to IMP administration.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to give written informed consent for participation in the study.
2. Healthy male or female subject aged ≥ 18 and ≤70 years.
3. Body Mass Index (BMI) ≥ 19.0 and ≤ 30.0 kg/m2.
4. Clinically normal medical history, physical findings, vital signs, ECG and laboratory values at the time of screening, as judged by the Investigator.
5. Women of child bearing potential (WOCBP) must practice abstinence from heterosexual intercourse (only allowed when this is the preferred and usual lifestyle of the subject) or must agree to use a highly effective method of contraception with a failure rate of < 1% to prevent pregnancy (combined [oestrogen and progestogen containing] hormonal contraception [oral, intravaginal, transdermal], progestogen-only hormonal contraception associated with inhibition of ovulation [oral, injectable, implantable], intrauterine device [IUD]or intrauterine hormone-releasing system [IUS]) from at least 4 weeks prior to dose to 4 weeks after last dose.

Exclusion Criteria:

1. Known allergy to GS-248.
2. Females who are breast feeding or who plan to become pregnant until 2 weeks after the end-of-study visit.
3. Positive serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) at screening and within 24 h prior to the first administration of IMP.
4. Regular use of corticosteroids (inhaled and systemic), NSAIDs, aspirin or coxibs, antacids, PPIs, or any other medication that changes gastric pH within 14 days of study drug administration.
5. Regular use of any prescribed or non-prescribed medication including analgesics, herbal remedies, vitamins and minerals within 2 weeks prior to the (first) administration of IMP, except hormonal contraception and occasional intake of paracetamol (maximum 2000 mg/day; and not exceeding 3000 mg/week) and nasal decongestants without cortisone, antihistamine or anticholinergics for a maximum of 10 days, at the discretion of the Investigator.
6. Presence of inherited or acquired disorders of platelet function, bleeding or coagulation, as judged by the investigator.
7. History or presence of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the subject at risk because of participation in the study, or influence the results or the subject's ability to participate in the study.
8. After 10 minutes supine rest at the time of screening, any vital signs values outside the following ranges:

   * Systolic blood pressure <90 or >140 mmHg, or
   * Diastolic blood pressure <50 or >90 mmHg, or
   * Pulse <40 or >90 bpm
9. Positive test for serum hepatitis B surface antigen (HBsAg), hepatitis C virus antibodies (HCVAb) or HIV 1 and/or 2 antibodies at screening.
10. Presence or history of drug and/or alcohol abuse and/or excessive intake of alcohol and/or history, or current use, of anabolic steroids, as judged by the Investigator.
11. Positive test for drugs of abuse or alcohol at screening or on admission to the unit prior to administration of the IMP.
12. Participation in other interventional studies within 3 months prior to administration of study drug.
13. Consumption of grapefruit, grapefruit juice, other grapefruit-containing products, or Seville oranges within 14 days of first IMP administration.
14. Any clinically significant illness, medical/surgical procedure or trauma within 4 weeks of the first administration of IMP.
15. Malignancy within the past 5 years with the exception of in situ removal of basal cell carcinoma.
16. Any planned major surgery within the duration of the study.
17. Prolonged QTcF (>450 ms), cardiac arrhythmias or any clinically significant abnormalities in the resting ECG, as judged by the Investigator.
18. Current smokers or users of nicotine products. Irregular use of nicotine (e.g., smoking, snuffing, chewing tobacco) less than three times per week is allowed before screening visit.
19. Regular excessive caffeine consumption defined by a daily intake of >5 cups of caffeine-containing beverages.
20. Intake of xanthine- and/or taurine-containing energy drinks within 2 days prior to screening and prior to IMP administration.
21. Plasma donation within one month of screening or blood donation (or corresponding blood loss) during three months prior to screening.
22. Investigator considers the subject unlikely to comply with study procedures, restrictions and requirements.
23. Estimated glomerular filtration rate (eGFR) < 50 mL/min/1.73 m2 (determined by the revised Lund-Malmö GFR estimating equation).
24. Subjects with swallowing disorders, which may affect the subject´s capability to swallow the IMP.
25. Subjects who are vegetarian or for other reasons cannot eat the high-fat high-calorie breakfast.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-03-31 (Actual); Primary Completion 2020-05-27 (Actual); Study Completion 2020-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Helena Litorp, MD, PhD, Principal Investigator — CTC Clinical Trial Consultants AB
Locations (1):
- Clinical Trial Consultants AB, Uppsala, Sweden

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The subjects were recruited from CTC's database of healthy volunteers and from advertising in media (including social media). Screening visits were performed at CTC research clinic.
  Recruitment period started 24MAR2020 (the day after approval received from IEC and CA) and lasted until 06APR2020 (date for last subject screened).
Pre-assignment Details: Screening (Visit 1) took place from Day -28 to Day -1 and included an eligibility check and a general health assessment. A total of 29 subjects were screened for participation. Eleven subjects were screening failures and 4 subjects were reserves who were not used in the study. Fourteen subjects were included and dosed in the study.
Groups:
- Part I GS-248 Formulation A: Formulation A given in fasting state.
  Formulation A GS-248: Formulation A of GS-248 in a lipid-based size 1 capsules, dose 120 mg given as a single-dose of 3 capsules a´40 mg.
- Part I GS-248 Formulation B: Formulation B given in fasting state.
  Formulation B GS-248: Formulation B of GS-248 in a dry powder size 1 capsules, dose 120 mg given as a single-dose of 3 capsules a´40 mg.
- Part II GS-248 Formulation A in Fed Condition: Formulation A given in fed condition. Formulation A was selected for the Food Interaction Part of the study, based on the PK profiles of both Formulation A and B.
  Formulation A of GS-248 in a capsule, dose 120 mg given as a single-dose of 3 capsules a´40 mg.
Period: Period 1: Part 1 Formulation A
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition
Started | 14 | 0 | 0 (Subjects were expected to participate in both Part I and Part II, seven visits in total. Subject 112 was prematurely withdrawn from the study due to self-reported Covid-19-like symptoms via phone after Visit 5, i.e. after receiving both GS-248 formulations but prior to the food interaction part. This means subject 112 was withdrawn after Part I Formulation B but before Part II which cannot be visualized in the Period section. The correct number of subjects started Part II is thus 13.)
Completed | 14 | 0 | 0
Not Completed | 0 | 0 | 0
Period: Period 2: Part 1 Formulation B
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition
Started | 0 | 14 | 0
Completed | 0 | 14 | 0
Not Completed | 0 | 0 | 0
Period: Period 3: Part 2 Formulation A Fed Cond.
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition
Started | 0 | 0 | 14
Completed | 0 | 0 | 13
Not Completed | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Overall Trial: All subjects who were included in the study i.e. randomized in Part I GS-248 Formulation A.
Arm/Group | Overall Trial
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.3 (17.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 13
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 14
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Sweden | 14
Height [Mean (Standard Deviation); unit: cm] | 171.6 (10.8)
Weight [Mean (Standard Deviation); unit: kg] | 74.5 (17.14)
BMI [Mean (Standard Deviation); unit: kg/m^2] | 25.1 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Cmax
Description: The Maximal Plasma Concentration (Cmax) after a single dose of Formulation A and B of GS 248 respectively in fasting conditions and after a single dose of Formulation A of GS-248 in fed condition.
  Blood samples for bioanalysis of GS-248 and subsequent PK analysis were collected as venous blood samples.
Time Frame: From time 0 (time of dosing) to 48 hours after dose (concentration measured at timepoints pre-dose and 0:15, 0:30, 1, 1:30, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: Part I Formulation A: Data based on Formulation PK analysis set i.e. 14 subjects.
  Part I Formulation B: Data based on Formulation PK analysis set i.e. 14 subjects.
  Part II Formulation A fed: Data based on Formulation PK analysis set i.e. 13 subjects.
  Part II Formulation A fasting (partial set): Data based on Formulation PK analysis set i.e. 13 subjects.
Measure: Mean (Standard Deviation); unit: nmol/L
Groups:
- Part II GS-248 Formulation A in Fed Condition: Formulation A given in fed condition. Formulation A was selected for the Food Interaction Part of the study, based on the PK profiles of both Formulation A and B.
  Formulation A of GS-248 in a capsule, dose 120 mg given as a single-dose of 3 capsules a´40 mg with breakfast.
- Part II GS-248 Formulation A in Fasting Condition (Partial Set): This arm (subject analysis set) was used for a comparison of PK parameters between Formulation A under fed and fasted conditions (namely calculation of the relative bioavailability). The analysis set is part of the Food Interaction PK Analysis Set (PKAS - Food Interaction), and consisted of all subjects in Arm 1 (receiving Formulation A under fasted conditions) who, subsequently, also received Formulation A under fed conditions in the third treatment period of the study (Arm 3). Since 1 subject terminated the study prematurely between study treatment period 1 and 3, only 13 subjects were included in this analysis set that was used for the assessment of the relative bioavailability of Formulation A in fed versus fasted conditions.
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition | Part II GS-248 Formulation A in Fasting Condition (Partial Set)
Number analyzed (Participants) | 14 | 14 | 13 | 13
nmol/L | 508.6 (220.9) | 384.5 (219.1) | 289.5 (184.4) | 499.5 (227.2)
Statistical Analysis 1: Comparison: Part I GS-248 Formulation A vs Part I GS-248 Formulation B vs Part II GS-248 Formulation A in Fasting Condition (Partial Set); Relative bioavailability (A versus B); Test type: Superiority — Relative bioavailability for Formulation A (FASTED) versus Formulation B (FASTED). The calculated relative bioavailability is based on Cmax ratio (ratio of geometric means) and is presented with 90% CI; Ratio of geometric means = 1.4514, 90% CI 2-sided [1.1110 to 1.4514]
Statistical Analysis 2: Comparison: Part II GS-248 Formulation A in Fed Condition vs Part II GS-248 Formulation A in Fasting Condition (Partial Set); Relative bioavailability (A FED versus A FASTED); Test type: Superiority — Relative bioavailability for Formulation A (FED) versus Formulation A (FASTED). The calculated relative bioavailability is based on Cmax ratio (ratio of geometric means) and is presented with 90% CI; Ratio of geometric mean = 0.5497, 90% CI 2-sided [0.3977 to 0.7597]

2. Primary Outcome: AUC0-inf
Description: The Area Under the Curve (AUC) for the time interval 0-infinity of GS-248 after a single dose of Formulation A and B of GS 248 respectively in fasting conditions and after a single dose of Formulation A of GS-248 in fed condition. The mean AUC of GS-248 was assessed by means of non-compartmental analysis (NCA).
  Blood samples for bioanalysis of GS-248 and subsequent PK analysis were collected as venous blood samples.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition | Part II GS-248 Formulation A in Fasting Condition (Partial Set)
Number analyzed (Participants) | 14 | 14 | 13 | 13
h*nmol/L | 1491 (478.1) | 1182 (567.4) | 1119 (463.9) | 1494 (497.4)
Statistical Analysis 1: Comparison: Part I GS-248 Formulation A vs Part I GS-248 Formulation B; Relative bioavailability (A versus B); Test type: Superiority — Relative bioavailability for Formulation A (FASTED) versus Formulation B (FASTED). The calculated relative bioavailability is based on AUC0-inf ratio (ratio of geometric means) and is presented with 90% CI; Ratio of geometric mean = 1.3441, 90% CI 2-sided [1.0953 to 1.6495]
Statistical Analysis 2: Comparison: Part II GS-248 Formulation A in Fed Condition vs Part II GS-248 Formulation A in Fasting Condition (Partial Set); Relative bioavailability (A FED versus A FASTED); Test type: Superiority — Relative bioavailability for Formulation A (FED) versus Formulation A (FASTED). The calculated relative bioavailability is based on AUC0-inf ratio (ratio of geometric means) and is presented with 90% CI; Ratio of geometric mean = 0.7327, 90% CI 2-sided [0.5910 to 0.9083]

3. Primary Outcome: AUC0-24h
Description: The Area Under the Curve (AUC) for the time interval 0-24h of GS-248 after a single dose of Formulation A and B of GS 248 respectively in fasting conditions and after a single dose of Formulation A of GS-248 in fed condition. The mean AUC of GS-248 for the time interval 0-24 h was assessed by means of non-compartmental analysis (NCA).
  Blood samples for bioanalysis of GS-248 and subsequent PK analysis were collected as venous blood samples.
Time Frame: From time 0 (time of dosing) to 24 hours after dose (concentration measured at timepoints pre-dose and 0:15, 0:30, 1, 1:30, 2, 3, 4, 6, 8, 12, 16, 24, 48 hours post-dose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h*nmol/L
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition | Part II GS-248 Formulation A in Fasting Condition (Partial Set)
Number analyzed (Participants) | 14 | 14 | 13 | 13
h*nmol/L | 1420 (459.4) | 1104 (527.2) | 1014 (377.6) | 1419 (478.2)
Statistical Analysis 1: Comparison: Part I GS-248 Formulation A vs Part I GS-248 Formulation B; Relative bioavailability (A versus B); Test type: Superiority — Relative bioavailability for Formulation A (FASTED) versus Formulation B (FASTED). The calculated relative bioavailability is based on AUC0-24h ratio (ratio of geometric means) and is presented with 90% CI; Ratio of geometric mean = 1.3710, 90% CI 2-sided [1.1120 to 1.6904]
Statistical Analysis 2: Comparison: Part II GS-248 Formulation A in Fed Condition vs Part II GS-248 Formulation A in Fasting Condition (Partial Set); Relative bioavailability (A FED versus A FASTED); Test type: Superiority — Relative bioavailability for Formulation A (FED) versus Formulation A (FASTED). The calculated relative bioavailability is based on AUC0-24h ratio (ratio of geometric means) and is presented with 90% CI; Ratio of geometric mean = 0.7083, 90% CI 2-sided [0.5728 to 0.8759]

4. Primary Outcome: Tmax
Description: Time to Cmax (Tmax) after a single dose of Formulation A and B of GS 248 respectively in fasting conditions and after a single dose of Formulation A of GS-248 in fed condition.
  Blood samples for bioanalysis of GS-248 and subsequent PK analysis were collected as venous blood samples.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hours
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition | Part II GS-248 Formulation A in Fasting Condition (Partial Set)
Number analyzed (Participants) | 14 | 14 | 13 | 13
hours | 1.500 [1.00 to 3.00] | 1.500 [1.00 to 3.03] | 3.000 [1.00 to 4.03] | 1.500 [1.00 to 3.00]

5. Primary Outcome: T1/2(z)
Description: Plasma half-life associated with the terminal elimination phase (T1/2(z)) after a single dose of Formulation A and B of GS 248 respectively in fasting conditions and after a single dose of Formulation A of GS-248 in fed condition.
  Blood samples for bioanalysis of GS-248 and subsequent PK analysis were collected as venous blood samples.
Time Frame: T1/2 (z) was assessed for the terminal elimination phase up to 48 hours
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition | Part II GS-248 Formulation A in Fasting Condition (Partial Set)
Number analyzed (Participants) | 14 | 14 | 13 | 13
hours | 10.69 (2.912) | 16.09 (15.26) | 13.36 (9.914) | 10.91 (2.902)

6. Primary Outcome: Vz/F
Description: The mean volume of distribution (Vz/F) after a single dose of Formulation A and B of GS 248 respectively in fasting conditions and after a single dose of Formulation A of GS-248 in fed condition.
  Blood samples for bioanalysis of GS-248 and subsequent PK analysis were collected as venous blood samples.
Time Frame: Vz/F was assessed for the terminal elimination phase up to 48 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition | Part II GS-248 Formulation A in Fasting Condition (Partial Set)
Number analyzed (Participants) | 14 | 14 | 13 | 13
L | 2071 (1035) | 3884 (2940) | 3110 (1588) | 2125 (1057)

7. Primary Outcome: CL/F
Description: The mean total clearance (CL/F) after a single dose of Formulation A and B of GS 248 respectively in fasting conditions and after a single dose of Formulation A of GS-248 in fed condition.
  The mean total clearance (CL/F) was calculated by non-compartmental analysis (NCA).
  Blood samples for bioanalysis of GS-248 and subsequent PK analysis were collected as venous blood samples.
Time Frame: CL/F was assessed for a single dose of GS-248 up to 48 hours.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/h
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition | Part II GS-248 Formulation A in Fasting Condition (Partial Set)
Number analyzed (Participants) | 14 | 14 | 13 | 13
L/h | 132.9 (50.59) | 191.4 (105.0) | 185.2 (76.08) | 133.7 (52.56)

8. Secondary Outcome: Number of Treatment Related Adverse Events
Description: The grading of the severity/intensity (grade 1 to grade 5) of AEs followed the common terminology criteria for AEs (CTCAE) v5.0. AEs were assessed by the Investigator as "unlikely", "possibly" or "probably" related to the IMP. An AE was considered causally related to the use of the IMP when the causality assessment was "probable" or "possible".
Time Frame: AEs (including serious AEs [SAEs]) were collected from the start of IMP application in Part I until the end-of- study visit i.e. Visit 7, day 3, up to 30 days.
Population: Part I Formulation A: Data based on safety analysis set i.e. 14 subjects. Part I Formulation B: Data based on safety analysis set i.e. 14 subjects. Part II Formulation A fed: Data based on safety analysis set i.e. 13 subjects.
Measure: Number; unit: events
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition
Number analyzed (Participants) | 14 | 14 | 13
events | 7 | 3 | 1

9. Secondary Outcome: Number of Clinically Significant (CS) Changes in Physical Examination
Description: A complete physical examination included assessments of the head, eyes, ears, nose, throat, skin, thyroid, neurological, lungs, cardiovascular, abdomen (liver and spleen), lymph nodes and extremities. A short version of physical examination included an assessment of selected body systems at the judgement of the Investigator but at least included cardiovascular, lung and abdomen.
  The results of the examinations were documented in the eCRF as normal, abnormal not clinically significant (NCS) or abnormal clinically significant (CS). Post-dose physical examination findings judged as abnormal CS were reported as AEs.
Time Frame: Physical examination was performed at pre-defined timepoints from the Screening Visit until the End-of- Study Visit i.e. Visit 7, day 3, up to 30 days.
Population: as for outcome 8
Measure: Number; unit: Number of abnormal CS events
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition
Number analyzed (Participants) | 14 | 14 | 13
Number of abnormal CS events | 0 | 0 | 0

10. Secondary Outcome: Number of Clinically Significant (CS) Changes in Vital Signs
Description: Systolic and diastolic blood pressure and pulse were measured in supine position after 10 minutes of rest. Vital signs were judged as normal, abnormal NCS or abnormal CS.
Time Frame: Vital signs ware assessed at pre-defined timepoints from the Screening Visit until the End-of- Study Visit i.e. Visit 7, day 3, up to 30 days.
Population: as for outcome 8
Measure: Number; unit: Number of abnormal CS events
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition
Number analyzed (Participants) | 14 | 14 | 13
Number of abnormal CS events | 0 | 0 | 0

11. Secondary Outcome: Number of Clinically Significant (CS) Changes in Resting 12-lead Electrocardiogram (ECG)
Description: Single 12-lead ECG was recorded in supine position after 10 minutes of rest using an ECG machine. HR and PR, QRS, QT and QTcF intervals were recorded. Safety ECGs were reviewed and interpreted on-site by the Investigator. All ECGs were categorised as "normal", "abnormal, not clinically significant", or "abnormal, clinically significant".
Time Frame: ECG evaluation was assessed at pre-defined timepoints from the Screening Visit until the End-of- Study Visit i.e. Visit 7, day 3, up to 30 days.
Population: as for outcome 8
Measure: Number; unit: Number of abnormal CS events
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition
Number analyzed (Participants) | 14 | 14 | 13
Number of abnormal CS events | 0 | 0 | 0

12. Secondary Outcome: Number of Clinically Significant (CS) Changes in Safety Laboratory Parameters
Description: Blood samples for analysis of clinical chemistry and haematology parameters were collected through venepuncture or an indwelling venous catheter and sent to the certified clinical chemistry laboratory at Uppsala University Hospital and analysed by routine analytical methods. Urine analysis was performed at the research clinic using dip sticks. Safety laboratory parameters were judged as normal, abnormal NCS or abnormal CS.
Time Frame: Blood samples were collected at pre-defined timepoints from the Screening Visit until the End-of- Study Visit i.e. Visit 7, day 3, up to 30 days.
Population: as for outcome 8
Measure: Number; unit: Number of abnormal CS events
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition
Number analyzed (Participants) | 14 | 14 | 13
Number of abnormal CS events | 0 | 1 | 1

ADVERSE EVENTS:
Time Frame: Adverse events, AEs (including SAEs), were collected from the start of IMP administration until the End-of-study Visit i.e. Visit 7, day 3, up to 30 days.
Description: The number of subjects that reported at least one adverse event (AE), or had at least one serious AE (SAE), including death, after administration of study product.
  The grading of the severity/intensity (grade 1 to grade 5) of AEs followed the common terminology criteria for AEs (CTCAE) v5.0. AEs were assessed as "unlikely", "possibly" or "probably" related to the IMP. An AE was considered causally related to the use of the IMP when the causality assessment was "probable" or "possible".
Arm/Group | Part I GS-248 Formulation A | Part I GS-248 Formulation B | Part II GS-248 Formulation A in Fed Condition
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/14 | 0/13
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 6/14 | 5/14 | 2/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part I GS-248 Formulation A (N=14) | Part I GS-248 Formulation B (N=14) | Part II GS-248 Formulation A in Fed Condition (N=13)
Headache (Nervous system disorders) | 6 (8) | 3 (3) | 1 (1) — Headache
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) — Anaemia
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) — Flatulence
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) — Haemoglobin decreased
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) — Rhinitis allergic

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any confidential information relating to the IMP or the study, including any data and results from the study, will be the exclusive property of the Sponsor. The Investigator and any other persons involved in the study are responsible for protecting the confidentiality of this proprietary information belonging to the Sponsor. The results from this study may be submitted for publication at the discretion of the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2020-01-29): https://cdn.clinicaltrials.gov/large-docs/09/NCT04617509/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-04): https://cdn.clinicaltrials.gov/large-docs/09/NCT04617509/SAP_001.pdf